CLINICAL TRIAL: NCT05977166
Title: Influence of Hyperbaric Oxygen on Pulmonary Functions in Post Covid-19 Patients.
Brief Title: Hyperbaric on Pulmonary Functions in Post Covid -19 Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Enas Faraman Mohamed, Physiothery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REL/012/003546
Record Dates: First submitted 2023-06-11; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Post COVID-19 Patients
MeSH Terms: interventions — Hyperbaric Oxygenation; Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyperbaric oxygen therapy ,breathing exercise,medical treatment (Active Comparator): Hyperbaric oxygen treatment HBO treatment was given daily in the morning on 21 consecutive days. (HBOT) treatment is a procedure performed inside a pressured chamber (the Hyperbaric Chamber). The patient is place inside the chamber exposure to 100% oxygen at 2 ATA with 5 min air breaks every 20 min. Each session consisted of 60 min. Measurements will be taken in the morning before entering, the first and last session.
  Interventions: Device: hyperbaric oxygen therapy; Device: breathing exercise; Drug: medical treatment
- breathing exercise and medical treatment (Active Comparator): breathing exercise completely each session of three repetitions initially. Every repetition consisted of one round of intervention 10-15 times followed by a brief rest (normal breathing) of <1 min (one repetition). Such 3 repetitions were given initially & advanced till 10 repetitions (one session) by last day of the week. In this manner participants practised 3 sessions twice a day, for a total duration of about 10-20 min every day.Vitamin D: The recommended dietary dose of vitamin D is 600 IU each day .
  Vitamine C: The recommended dietary dose 200 mg/day vitamin C. Anticoagulation drugs (blood thinners), doctors usually prescribe low-molecular-weight heparin (enoxaparin) (30 mg), each given subcutaneously every 12 hours
  Interventions: Device: hyperbaric oxygen therapy; Device: breathing exercise; Drug: medical treatment

INTERVENTIONS:
Device: hyperbaric oxygen therapy — All patients participated in the current study will receive breathing excesses in form of Diaphragmatic breathing exercise and Pursed lip breathing with traditional medical treatment in form of (vitamin D, vitamin C and Anticoagulation drugs ,group A will receive 60 minutes of HBOT(100%oxygen at 2 ATA with five minutes air breaks every twenty minutes daily in morning for three weeks then take period time of rest about 30 minutes before starting breathing exercise.
Device: breathing exercise — All patients participated in the current study will receive breathing excesses in form of Diaphragmatic breathing exercise and Pursed lip breathing with traditional medical treatment in form of (vitamin D, vitamin C and Anticoagulation drugs ,group A will receive 60 minutes of HBOT(100%oxygen at 2 ATA with five minutes air breaks every twenty minutes daily in morning for three weeks then take period time of rest about 30 minutes before starting breathing exercise.
Drug: medical treatment — All patients participated in the current study will receive breathing excesses in form of Diaphragmatic breathing exercise and Pursed lip breathing with traditional medical treatment in form of (vitamin D, vitamin C and Anticoagulation drugs ,group A will receive 60 minutes of HBOT(100%oxygen at 2 ATA with five minutes air breaks every twenty minutes daily in morning for three weeks then take period time of rest about 30 minutes before starting breathing exercise.

SUMMARY:
Purpose of the study is to investigate the effect of hyperbaric oxygen on FVC, FEV1 and on oxygen saturation in post-COVID-19 patients, The effect of breathing exercises in form of diaphragmatic breathing exercise and pursed lip breathing with traditional medical treatment in form of (vitamin D, vitamin C and anticoagulation drugs on FVC, FEV1 and on oxygen saturation in post-COVID-19 patients.and the difference between the effect of hyperbaric and breathing exercises in form of diaphragmatic breathing exercise and pursed lip breathing with traditional medical treatment in form of (vitamin D, vitamin C and anticoagulation drugs on FVC, FEV1 and on oxygen saturation in post-COVID-19 patients

Seventy two covid-19 patients from both genders ranged in age chronology from twenty one to sixty six years will be conducted to participate in this study .Selection of the study sample and evaluate of pulmonary functions improvement as well as hyperbaric oxygen therapy will be conducted at Agriculture Hospital in El Mansoura town.

The study sample will be divided randomly into two equal groups of(A&B).All patients participated in the current study will receive breathing excesses in form of Diaphragmatic breathing exercise and Pursed lip breathing with traditional medical treatment in form of (vitamin D, vitamin C and Anticoagulation drugs ,group A will receive 60 minutes of HBOT(100%oxygen at 2 ATA with five minutes air breaks every twenty minutes daily in morning for three weeks then take period time of rest about 30 minutes before starting breathing exercise.

The Body mass index (BMI) of each participated patient will be determined by measuring weight/ Kg and height/ m2 using Electronic weight and height scale to include BMI 25.0-29.9 Kg/ . Also using Digital spirometer SMP 21/01 RD (Russian) for measuring of FVC parameters , to be less than 80% ,FEV1 to be less than 80% and Pulse Oximeter for measuring Oxygen saturation to range from 90%to 95% assessment will be done before and after treatment.

The obtained results of this study will measure Forced vital capacity (FVC), Forced expiratory volume (FEV1) and oxygen saturation to determine the significant improvement of participated patients.

ELIGIBILITY:
Inclusion Criteria

* 1. post Covid -19 patients (2weeks after recovery).

  2.post Covid -19 patients with deficiency in forced vital capacity (less than 80%) forced expiratory volume (less than 80%) lower oxygen saturation (90%-95%).

  3.age (21-66)years old.

  4.both gender.

  5.BMI 25.0-29.9.

Exclusion Criteria:

1. COPD or other respiratory diseases.
2. Neurological disease.
3. mental illness.
4. Critically ill patients with intubation.
5. smokers.
6. Inner ear diseases.
7. pregnancy.

Ages: 21 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
forced vital capacity, | 3 Months
  by spirometer
forced expiratory volume | 3 Months
  by spirometer
oxygen saturation | 3 Months
  pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Enas Faraman, Principal Investigator — physiothyrapist at kafer Elshikh general Hospital
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No